CLINICAL TRIAL: NCT05691478
Title: A Feasibility and Randomized Phase 2/3 Study of the VEGFR2/MET Inhibitor Cabozantinib in Combination With Cytotoxic Chemotherapy for Newly Diagnosed Osteosarcoma
Brief Title: A Study to Test the Addition of the Drug Cabozantinib to Chemotherapy in Patients With Newly Diagnosed Osteosarcoma
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2022-08567; NCI-2022-08567 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AOST2032 (Other: Children's Oncology Group); AOST2032 (Other: CTEP); U10CA180886 (NIH); NCT05683197 (obsolete NCT alias)
Record Dates: First submitted 2023-01-18; First posted 2023-01-20 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-09

CONDITIONS: High Grade Osteosarcoma; Localized Osteosarcoma; Metastatic Osteosarcoma; Secondary Osteosarcoma
MeSH Terms: conditions — Osteosarcoma | interventions — cabozantinib; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Doxorubicin; Magnetic Resonance Spectroscopy; Methotrexate; merphos; Surgical Procedures, Operative; X-Rays; Phantoms, Imaging

STUDY DESIGN:
Intervention Model Description: Single-arm Feasibility Phase study followed by a randomized, parallel 4-arm Efficacy Phase study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Efficacy Phase Arm A (MAP) (Active Comparator): Standard risk patients receive methotrexate IV, doxorubicin IV, and cisplatin IV for two 35-day "induction" cycles, followed by appropriate local control. Patients then receive "consolidation" with methotrexate IV, doxorubicin IV, and cisplatin IV for two 35-day cycles and methotrexate IV and doxorubicin IV for two additional 35-day cycles. Patients also undergo X-ray, CT, MRI, and PET or bone scintigraphy at diagnosis and additional time points throughout the trial. All patients also undergo collection of blood samples during screening and on study.
  Interventions: Procedure: Bone Scan; Drug: Cisplatin; Procedure: Computed Tomography; Drug: Doxorubicin Hydrochloride; Procedure: Magnetic Resonance Imaging; Drug: Methotrexate; Procedure: Surgical Procedure; Procedure: X-Ray Imaging
- Efficacy Phase Arm B (cabozantinib, MAP) (Experimental): Standard risk patients receive cabozantinib PO, methotrexate IV, doxorubicin IV, and cisplatin IV for two 35-day "induction" cycles, followed by appropriate local control. Patients then receive one 35-day "consolidation" cycle with methotrexate IV, doxorubicin IV, and cisplatin IV, then a second 35-day "consolidation" cycle with cabozantinib PO, methotrexate IV, doxorubicin IV, and cisplatin IV, followed by two additional 35-day "consolidation" cycles with cabozantinib PO, methotrexate IV, and doxorubicin IV. Patients then receive cabozantinib PO for six 28-day "maintenance" cycles. Patients also undergo X-ray, CT, MRI, and PET or bone scintigraphy at diagnosis and additional time points throughout the trial. All patients also undergo collection of blood samples during screening and on study.
  Interventions: Procedure: Bone Scan; Drug: Cabozantinib S-malate; Drug: Cisplatin; Procedure: Computed Tomography; Drug: Doxorubicin Hydrochloride; Procedure: Magnetic Resonance Imaging; Drug: Methotrexate; Procedure: Surgical Procedure; Procedure: X-Ray Imaging
- Efficacy Phase Arm C (MAP) (Active Comparator): High risk patients receive methotrexate IV, doxorubicin IV, and cisplatin IV for two 35-day "induction" cycles, followed by appropriate local control. Patients then receive "consolidation" with methotrexate IV, doxorubicin IV, and cisplatin IV for two 35-day cycles and methotrexate IV and doxorubicin IV for two additional 35-day cycles. Patients also undergo X-ray, CT, MRI, and PET or bone scintigraphy at diagnosis and additional time points throughout the trial. All patients also undergo collection of blood samples during screening and on study.
  Interventions: Procedure: Bone Scan; Drug: Cisplatin; Procedure: Computed Tomography; Drug: Doxorubicin Hydrochloride; Procedure: Magnetic Resonance Imaging; Drug: Methotrexate; Procedure: Surgical Procedure; Procedure: X-Ray Imaging
- Efficacy Phase Arm D (cabozantinib, MAP) (Experimental): High risk patients receive cabozantinib PO, methotrexate IV, doxorubicin IV, and cisplatin IV for two 35-day "induction" cycles, followed by appropriate local control. Patients then receive one 35-day "consolidation" cycle with methotrexate IV, doxorubicin IV, and cisplatin IV, then a second 35-day "consolidation" cycle with cabozantinib PO, methotrexate IV, doxorubicin IV, and cisplatin IV, followed by two additional 35-day "consolidation" cycles with cabozantinib PO, methotrexate IV, and doxorubicin IV. Patients then receive cabozantinib PO for six 28-day "maintenance" cycles. Patients also undergo X-ray, CT, MRI, and PET or bone scintigraphy at diagnosis and additional time points throughout the trial. All patients also undergo collection of blood samples during screening and on study.
  Interventions: Procedure: Bone Scan; Drug: Cabozantinib S-malate; Drug: Cisplatin; Procedure: Computed Tomography; Drug: Doxorubicin Hydrochloride; Procedure: Magnetic Resonance Imaging; Drug: Methotrexate; Procedure: X-Ray Imaging
- Feasibility phase (cabozantinib, MAP) (Experimental): (CLOSED TO ACCRUAL 05/09/2025): Patients receive cabozantinib orally (PO), methotrexate intravenously (IV), doxorubicin IV, and cisplatin IV for two 35-day "induction" cycles. Patients are then considered for appropriate local control. Then they receive "consolidation" with methotrexate IV, doxorubicin IV, and cisplatin IV for one 35-day cycle, followed by cabozantinib PO, methotrexate IV, doxorubicin IV, and cisplatin IV for one 35-day cycle, and cabozantinib PO, methotrexate IV, and doxorubicin IV for two 35-day cycles. Patients then receive cabozantinib PO for six 28-day "maintenance" cycles.
  Interventions: Procedure: Bone Scan; Drug: Cabozantinib S-malate; Drug: Cisplatin; Procedure: Computed Tomography; Drug: Doxorubicin Hydrochloride; Procedure: Magnetic Resonance Imaging; Drug: Methotrexate; Procedure: Surgical Procedure; Procedure: X-Ray Imaging

INTERVENTIONS:
Procedure: Bone Scan — Undergo bone scintography
  Other Names: Bone Scintigraphy
Drug: Cabozantinib S-malate — Given PO
  Other Names: BMS-907351; Cabometyx; Cometriq; XL 184; XL-184; XL184
  Arms: Efficacy Phase Arm B (cabozantinib, MAP); Efficacy Phase Arm D (cabozantinib, MAP); Feasibility phase (cabozantinib, MAP)
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; FI106; hydroxydaunorubicin; Rubex
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Methotrexate — Given IV
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Jylamvo; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Procedure: Surgical Procedure — Undergo surgery
  Other Names: Operation; Surgery; Surgery Type; Surgery, NOS; Surgical; Surgical Intervention; Surgical Interventions; Surgical Procedures; Type of Surgery
  Arms: Efficacy Phase Arm A (MAP); Efficacy Phase Arm B (cabozantinib, MAP); Efficacy Phase Arm C (MAP); Feasibility phase (cabozantinib, MAP)
Procedure: X-Ray Imaging — Undergo X-ray
  Other Names: Conventional X-Ray; Diagnostic Radiology; Medical Imaging, X-Ray; Plain film radiographs; Radiographic Imaging; Radiographic imaging procedure (procedure); Radiography; RG; Static X-Ray; X-Ray

SUMMARY:
This phase II/III trial tests the safety, side effects, and best dose of the drug cabozantinib in combination with standard chemotherapy, and to compare the effect of adding cabozantinib to standard chemotherapy alone in treating patients with newly diagnosed osteosarcoma. Cabozantinib is in a class of medications called kinase inhibitors which block protein signals affecting new blood vessel formation and the ability to activate growth signaling pathways. This may help slow the growth of tumor cells. The drugs used in standard chemotherapy for this trial are methotrexate, doxorubicin, and cisplatin (MAP). Methotrexate stops cells from making DNA and may kill tumor cells. It is a type of antimetabolite. Doxorubicin is in a class of medications called anthracyclines. It works by slowing or stopping the growth of tumor cells in the body. Cisplatin is in a class of medications known as platinum-containing compounds. It works by killing, stopping or slowing the growth of tumor cells. Adding cabozantinib to standard chemotherapy may work better in treating newly diagnosed osteosarcoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility of adding cabozantinib S-malate (cabozantinib) to standard MAP (high dose methotrexate, doxorubicin hydrochloride [doxorubicin], and cisplatin) chemotherapy in patients with newly diagnosed metastatic osteosarcoma with a resectable primary tumor.

II. To determine whether MAP chemotherapy plus cabozantinib results in more favorable event-free survival (EFS) than MAP chemotherapy alone in patients with localized, resectable osteosarcoma.

III. To determine whether MAP chemotherapy plus cabozantinib results in more favorable event-free survival (EFS) than MAP chemotherapy alone in patients with metastatic, pelvic and unresectable osteosarcoma.

SECONDARY OBJECTIVES:

I. To determine whether MAP chemotherapy plus cabozantinib results in more favorable overall survival (OS) than MAP chemotherapy alone in patients with localized, resectable osteosarcoma.

II. To determine whether MAP chemotherapy plus cabozantinib results in more favorable overall survival (OS) than MAP chemotherapy alone in patients with metastatic, pelvic and unresectable osteosarcoma.

III. To prospectively validate that elevated circulating tumor DNA (ctDNA) levels greater than or equal to 5% at the time of diagnosis are associated with increased risk of EFS-event in patients with localized, resectable osteosarcoma.

IV. To prospectively validate that elevated ctDNA levels greater than or equal to 5% at the time of diagnosis are associated with increased risk of EFS-event in patients with metastatic, pelvic and unresectable osteosarcoma.

V. To prospectively validate that elevated ctDNA levels greater than or equal to 3% after initiation of therapy and prior to definitive surgery are associated with increased risk of EFS-event in patients with localized, resectable osteosarcoma.

VI. To prospectively validate that elevated ctDNA levels greater than or equal to 3% after initiation of therapy and prior to definitive surgery are associated with increased risk of EFS-event in patients with metastatic, pelvic and unresectable osteosarcoma.

VII. To determine whether MAP chemotherapy plus cabozantinib results in increased symptom burden and decreased tolerability to patients as measured by patient reported therapy-specific acute toxicities (Patient-Reported Outcomes-Common Terminology Criteria for Adverse Events [PRO-CTCAE]).

EXPLORATORY OBJECTIVES:

I. To determine the rate of good histologic response (> 90%) of resected primary tumor specimens following neoadjuvant chemotherapy with MAP plus cabozantinib and compare with response rates for MAP chemotherapy alone.

II. To describe the toxicities of the addition of cabozantinib to MAP chemotherapy in patients with newly diagnosed osteosarcoma.

III. To compare the probability of Grade 3 or higher port site wound complications on the MAP plus cabozantinib regimen to that of MAP chemotherapy alone in patients with newly diagnosed osteosarcoma who received a port for the administration of chemotherapy.

IV. To describe frequency of application of local control methods (surgery, hypofractionated stereotactic body radiotherapy, or radiofrequency ablation) for extrapulmonary metastatic osteosarcoma.

V. To compare total cumulative delivered doses of MAP chemotherapy agents between standard and experimental arms across multiple phases of therapy.

VI. To assess the pharmacokinetics of cabozantinib when administered concomitantly with standard chemotherapy agents during feasibility.

VII. To collect pulmonary metastatic lesions, paired primary tumor tissue, and serial blood samples for tumor profiling, liquid biopsies, and future testing of correlative biology studies.

VIII. To determine whether ctDNA at diagnosis and early on-treatment, as a continuous measurement of ctDNA burden, is associated with an increased risk of EFS-event in patients with newly diagnosed osteosarcoma.

IX. To evaluate whether the magnitude of change in ctDNA levels from diagnosis to planned surgical procedure is associated with risk of EFS-event in patients with newly diagnosed osteosarcoma.

X. To determine whether ctDNA levels greater than or equal to 3% after planned surgical procedures are associated with increased risk of EFS-event.

XI. To describe the presence of specific copy-number alterations, including MYC amplifications, detected in ctDNA and matched diagnostic tumor samples in patients with newly diagnosed osteosarcoma and determine whether frequently occurring copy-number alterations are associated with increased risk of EFS-event.

XII. To determine whether ctDNA burden is predictive of response to the experimental therapy in patients with newly diagnosed osteosarcoma.

XIII. To prospectively compare the impact of combination therapy on symptom bother as measured by the Functional Assessment of Cancer Therapy-General Questionnaire (FACT-G) item GP5 in patients with osteosarcoma receiving MAP chemotherapy with or without cabozantinib, and to assess the relationship between symptom bother and number of patient-reported acute toxicities (as measured by the PRO-CTCAE).

OUTLINE: This is a dose-escalation study of cabozantinib (Feasibility Phase) followed by a randomized phase II/III study (Efficacy Phase).

FEASIBILITY PHASE (CLOSED TO ACCRUAL 05/09/2025): Patients receive cabozantinib orally (PO), methotrexate intravenously (IV), doxorubicin IV, and cisplatin IV for two 35-day "induction" cycles. Patients are then considered for appropriate local control. Then they receive "consolidation" with methotrexate IV, doxorubicin IV, and cisplatin IV for one 35-day cycle, followed by cabozantinib PO, methotrexate IV, doxorubicin IV, and cisplatin IV for one 35-day cycle, and cabozantinib PO, methotrexate IV, and doxorubicin IV for two 35-day cycles. Patients then receive cabozantinib PO for six 28-day "maintenance" cycles.

EFFICACY PHASE: Patients with standard risk osteosarcoma are randomized to Arm A or Arm B. Patients with high risk osteosarcoma are randomized to Arm C or Arm D.

ARM A: Standard risk patients receive methotrexate IV, doxorubicin IV, and cisplatin IV for two 35-day "induction" cycles, followed by appropriate local control. Patients then receive "consolidation" with methotrexate IV, doxorubicin IV, and cisplatin IV for two 35-day cycles and methotrexate IV and doxorubicin IV for two additional 35-day cycles.

ARM B: Standard risk patients receive cabozantinib PO, methotrexate IV, doxorubicin IV, and cisplatin IV for two 35-day "induction" cycles, followed by appropriate local control. Patients then receive one 35-day "consolidation" cycle with methotrexate IV, doxorubicin IV, and cisplatin IV, then a second 35-day "consolidation" cycle with cabozantinib PO, methotrexate IV, doxorubicin IV, and cisplatin IV, followed by two additional 35-day "consolidation" cycles with cabozantinib PO, methotrexate IV, and doxorubicin IV. Patients then receive cabozantinib PO for six 28-day "maintenance" cycles.

ARM C: High risk patients receive methotrexate IV, doxorubicin IV, and cisplatin IV for two 35-day "induction" cycles, followed by appropriate local control. Patients then receive "consolidation" with methotrexate IV, doxorubicin IV, and cisplatin IV for two 35-day cycles and methotrexate IV and doxorubicin IV for two additional 35-day cycles.

ARM D: High risk patients receive cabozantinib PO, methotrexate IV, doxorubicin IV, and cisplatin IV for two 35-day "induction" cycles, followed by appropriate local control. Patients then receive one 35-day "consolidation" cycle with methotrexate IV, doxorubicin IV, and cisplatin IV, then a second 35-day "consolidation" cycle with cabozantinib PO, methotrexate IV, doxorubicin IV, and cisplatin IV, followed by two additional 35-day "consolidation" cycles with cabozantinib PO, methotrexate IV, and doxorubicin IV. Patients then receive cabozantinib PO for six 28-day "maintenance" cycles.

All patients also undergo X-ray, computed tomography (CT), magnetic resonance imaging (MRI), and positron emission tomography (PET) or bone scintigraphy at diagnosis and additional time points throughout the trial. All patients also undergo collection of blood samples during screening and on study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be < 40 years of age at the time of enrollment.
* Patients must have a body surface area of >= 0.8 m^2 at the time of enrollment.
* Patients must have histologic diagnosis (by institutional pathologist) of newly diagnosed high grade osteosarcoma. Primary tumors of all extremity and axial sites are eligible as long as diagnosis of high-grade osteosarcoma is established. Osteosarcoma as a second malignancy is eligible if no prior exposure to systemic chemotherapies.
* Feasibility Phase (NOTE: as of Amendment #2B, the feasibility phase has been completed) Patients must have metastatic disease and a resectable primary tumor. Designation of a primary tumor as resectable will be determined at the time of diagnosis by the institutional multidisciplinary team.

For this study, metastatic disease is defined as one or more of the following:

* Lesions which are discontinuous from the primary tumor, are not regional lymph nodes, and do not share a bone or body cavity with the primary tumor. Skip lesions in the same bone as the primary tumor do not constitute metastatic disease. Skip lesions in an adjacent bone are considered bone metastases.
* Lung metastases: defined as biopsy-proven metastasis or the presence of one or more pulmonary lesions >= 5 mm, OR multiple pulmonary lesions >= 3 mm or greater in size.
* Bone metastases: Areas suspicious for bone metastasis based on fludeoxyglucose F-18 (18F-FDG)-positron emission tomography (PET) scan (or whole body technetium-99 bone scan if 18F-FDG-PET is unavailable at the treating institution) require confirmatory biopsy or supportive anatomic imaging of at least one suspicious site with either magnetic resonance imaging (MRI) or computed tomography (CT) (whole body 18F-FDG-PET/CT or 18F-FDG-PET/MR scans are acceptable).

  * Efficacy Phases (Phase 2/3) NOTE: as of Amendment #2B, the efficacy phase is open for enrollment.

Patients with both localized and metastatic disease are eligible for the efficacy phase, regardless of resectability. Patients will be enrolled to two separate cohorts:

* Cohort 1 (Standard Risk): Patients with non-pelvic primary osteosarcoma deemed to be resectable at the time of diagnosis by the institutional multidisciplinary team, without evidence of metastatic lesions.
* Cohort 2 (High-Risk): Patients with a primary pelvic tumor, a primary tumor designated as unresectable by the institutional multidisciplinary team, AND/OR radiographic evidence of metastatic lesions.

  * A serum creatinine based on age/sex as follows (within 7 days prior to enrollment unless otherwise indicated):
* (Age: Maximum Serum Creatinine [mg/dL]; Sex)

  * 1 month to < 6 months: 0.4 (male); 0.4 (female)
  * 6 months to < 1 year: 0.5 (male); 0.5 (female)
  * 1 to < 2 years: 0.6 (male); 0.6 (female)
  * 2 to < 6 years: 0.8 (male); 0.8 (female)
  * 6 to < 10 years: 1 (male); 1 (female)
  * 10 to < 13 years: 1.2 (male); 1.2 (female)
  * 13 to < 16 years: 1.5 (male); 1.4 (female)
  * >= 16 years: 1.7 (male); 1.4 (female)
* OR - a 24 hour urine creatinine clearance >= 70 mL/min/1.73 m^2
* OR - a glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2. GFR must be performed using direct measurement with a nuclear blood sampling method OR direct small molecule clearance method (iothalamate or other molecule per institutional standard).

  * Note: Estimated GFR (eGFR) from serum creatinine, cystatin C or other estimates are not acceptable for determining eligibility.

    * Total bilirubin =< 1.5 x upper limit of normal (ULN) for age (within 7 days prior to enrollment unless otherwise indicated)
    * Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 135 U/L (within 7 days prior to enrollment unless otherwise indicated)
* Note: For the purpose of this study, the ULN for SGPT (ALT) has been set to the value of 45 U/L

  * No history of congenital prolonged corrected QT (QTc) syndrome, New York Heart Association (NYHA) Class III or IV congestive heart failure, unstable angina pectoris, serious cardiac arrhythmias
* Shortening fraction of >= 27%, or
* Ejection fraction of >= 50%
* Corrected QT interval by Fridericia (QTcF) < 480 msec on electrocardiogram. Patients with Grade 1 prolonged QTc (450-480 msec) at time of study enrollment should have correctable causes of prolonged QTc addressed if possible (i.e., electrolytes, medications).

  * Peripheral absolute neutrophil count (ANC) >= 1000/uL (within 7 days prior to enrollment unless otherwise indicated)
  * Platelet count >= 100,000/uL (transfusion independent, defined as not receiving platelet transfusions within a 7-day period prior to enrollment) (within 7 days prior to enrollment unless otherwise indicated)
  * Hemoglobin >= 8.0 g/dL (within 7 days prior to enrollment unless otherwise indicated)
  * International normalized ratio (INR) =< 1.5 (within 7 days prior to enrollment unless otherwise indicated)
  * Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible as long as they are NOT receiving anti-retroviral agents that are strong inhibitors or inducers of CYP3A4, CYP2D6, and/or MRP2 transporter protein.
  * All patients and/or their parents or legal guardians must sign a written informed consent.
  * All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met.

Exclusion Criteria:

* Patients who have received previous systemic therapy for osteosarcoma or a prior oncologic diagnosis.
* Patients who have central nervous system metastases.
* Patients with central cavitating pulmonary lesions invading or encasing any major blood vessels in the lung.
* Patients who are unable to swallow tablets. Tablets cannot be crushed or chewed.
* Patients with gastrointestinal disorders including active disorders associated with a high risk of perforation or fistula formation. Specifically, no clinically significant gastrointestinal (GI) bleeding, GI perforation, bowel obstruction, intra-abdominal abscess or fistula for 6 months prior to enrollment, no hemoptysis or other signs of pulmonary hemorrhage for 3 months prior to enrollment.
* Patients with active bleeding or bleeding diathesis. No clinically significant hematuria, hematemesis, or hemoptysis or other history of significant bleeding within 3 months prior to enrollment.
* Patients with uncompensated or symptomatic hypothyroidism. Patients who have hypothyroidism controlled with thyroid replacement hormone are eligible.
* Patients with moderate to severe hepatic impairment (Child-Pugh B or C).
* Patients who have had primary tumor resection or attempted curative resection of metastases prior to enrollment.
* Patients who have undergone other major surgical procedure (eg, laparotomy) within 14 days prior to enrollment. Thoracoscopic procedures for diagnostic purposes (biopsy of lung nodule) and central access such as port-a-cath placement are allowed.
* Patients with a history of serious or non-healing wound or bone fracture (pathologic fracture of primary tumor is not considered exclusion).
* Patients with any medical or surgical conditions that would interfere with gastrointestinal absorption of cabozantinib.
* Patients with previously identify allergy or hypersensitivity to components of the study treatment formulations.
* Patients who are receiving any other investigational agent not defined within this protocol are not eligible.
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible.
* Patients who received enzyme-inducing anticonvulsants within 14 days prior to enrollment.
* Patients with a prior history of hypertension (> 95th percentile for age, height, and sex for patients < 18 years and > 140/90 mmHg for patients >= 18 years requiring medication for blood pressure control.
* Patients who are receiving drugs that prolong QTc.
* Patients receiving anticoagulation with oral coumarin agents (eg warfarin), direct thrombin inhibitors (eg dabigatran), direct factor Xa inhibitor betrixaban, or platelet inhibitors (eg, clopidogrel). Low dose aspirin for cardioprotection (per local applicable guidelines) and low dose, low molecular weight heparins (LMWH) are permitted. Anticoagulation with therapeutic doses of LMWH and direct factor Xa inhibitors rivaroxaban or apixaban are allowed in subjects who are on a stable dose for at least 6 weeks before the first dose of study treatment, and who have had no complications from a thromboembolic event or the anticoagulation regimen.
* Patients receiving strong CYP3A4 inducers or strong CYP3A4 inhibitors.
* Female patients who are pregnant since fetal toxicities and teratogenic effects have been noted for several of the study drugs. A pregnancy test is required for female patients of childbearing potential.
* Lactating females who plan to breastfeed their infants.
* Sexually active patients of reproductive potential who have not agreed to use an effective contraceptive method for the duration of protocol therapy.

Max Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1122 (Estimated)
Dates: Start 2023-03-03 (Actual); Primary Completion 2030-03-20 (Estimated); Study Completion 2030-03-20 (Estimated)

PRIMARY OUTCOMES:
Occurrence of dose-limiting toxicity (Feasibility) | Baseline up to 6 weeks
  Only patients with high risk osteosarcoma who have a primary tumor considered resectable at the time of enrollment will be enrolled to this part of the trial. If a feasible dose cannot be established, the study committee will consult with Children's Oncology Group leadership and National Cancer Institute Cancer Therapy Evaluation Program regarding possible modifications of the regimen and subsequent protocol amendment.
Event-free survival (EFS) (Phase II) | From randomization until disease progression, relapse, diagnosis of a second malignant neoplasm, death or last contact, whichever occurs first, assessed up to 5 years after completion of study treatment
  The randomization and analysis will be stratified according to risk group. An assessment of the reduction in risk for EFS-event at the designated landmark time will be used to determine whether the trial continues to part 3. If the study proceeds to part 3, patients enrolled to part 2 of the trial will contribute to the primary analyses for part 3 of the study. If the interim criterion for continuation is not obtained, accrual will be closed with the conclusion that cabozantinib does not reduce sufficiently the risk for EFS-event for patients with newly-diagnosed osteosarcoma.
EFS (Phase III) | From randomization until disease progression, relapse, diagnosis of a second malignant neoplasm, death or last contact, whichever occurs first, assessed up to 5 years after completion of study treatment
  Will consist of two randomized phase 3 sub-studies ('Phase 3'). One will be conducted in standard risk patients and one will be conducted in high risk patients.
Overall survival | From randomization until death or last contact, whichever occurs first, assessed up to 5 years after completion of study treatment

SECONDARY OUTCOMES:
EFS | From randomization until disease progression, relapse, diagnosis of a second malignant neoplasm, death or last contact, whichever occurs first, assessed up to 5 years after completion of study treatment
  Will validate whether elevated circulating tumor deoxyribonucleic acid (ctDNA) levels greater than or equal to 5% at the time of diagnosis are associated with increased risk of EFS-event in patients with localized, resectable osteosarcoma.
EFS | From randomization until disease progression, relapse, diagnosis of a second malignant neoplasm, death or last contact, whichever occurs first, assessed up to 5 years after completion of study treatment
  Will validate whether elevated ctDNA levels greater than or equal to 5% at the time of diagnosis are associated with increased risk of EFS-event in patients with metastatic, pelvic and unresectable osteosarcoma.
EFS | From randomization until disease progression, relapse, diagnosis of a second malignant neoplasm, death or last contact, whichever occurs first, assessed up to 5 years after completion of study treatment
  Will validate whether elevated ctDNA levels greater than or equal to 3% after initiation of therapy and prior to definitive surgery are associated with increased risk of EFS-event in patients with localized, resectable osteosarcoma.
EFS | From randomization until disease progression, relapse, diagnosis of a second malignant neoplasm, death or last contact, whichever occurs first, assessed up to 5 years after completion of study treatment
  Will validate whether elevated ctDNA levels greater than or equal to 3% after initiation of therapy and prior to definitive surgery are associated with increased risk of EFS-event in patients with metastatic, pelvic and unresectable osteosarcoma.
Change in symptom burden and tolerability | Up to 5 years after completion of study treatment
  Will determine whether methotrexate, doxorubicin, and cisplatin (MAP) chemotherapy plus cabozantinib results in increased symptom burden and decreased tolerability to patients as measured by patient reported therapy-specific acute toxicities (Patient-Reported Outcomes-Common Terminology Criteria for Adverse Events [PRO-CTCAE]).

OTHER OUTCOMES:
EFS | From randomization until disease progression, relapse, diagnosis of a second malignant neoplasm, death or last contact, whichever occurs first, assessed up to 5 years after completion of study treatment
  Will determine whether ctDNA at diagnosis and early on-treatment, as a continuous measurement of ctDNA burden, is associated with an increased risk of EFS-event in patients with newly diagnosed osteosarcoma.
EFS | From randomization until disease progression, relapse, diagnosis of a second malignant neoplasm, death or last contact, whichever occurs first, assessed up to 5 years after completion of study treatment
  Will evaluate whether the magnitude of change in ctDNA levels from diagnosis to planned surgical procedure is associated with risk of EFS-event in patients with newly diagnosed osteosarcoma.
EFS | From randomization until disease progression, relapse, diagnosis of a second malignant neoplasm, death or last contact, whichever occurs first, assessed up to 5 years after completion of study treatment
  Will determine whether ctDNA levels greater than or equal to 3% after planned surgical procedures are associated with increased risk of EFS-event.
EFS | From randomization until disease progression, relapse, diagnosis of a second malignant neoplasm, death or last contact, whichever occurs first, assessed up to 5 years after completion of study treatment
  Will describe the presence of specific copy-number alterations, including MYC amplifications, detected in ctDNA and matched diagnostic tumor samples in patients with newly diagnosed osteosarcoma and determine whether frequently occurring copy-number alterations are associated with increased risk of EFS-event.
ctDNA burden | Up to 5 years after completion of study treatment
  Will determine whether ctDNA burden is predictive of response to the experimental therapy in patients with newly diagnosed osteosarcoma.
Impact of combination therapy on symptom bother | Up to 5 years after completion of study treatment
  Will prospectively compare the impact of combination therapy on symptom bother as measured by the Functional Assessment of Cancer Therapy-General Questionnaire item GP5 in patients with osteosarcoma receiving MAP chemotherapy with or without cabozantinib, and to assess the relationship between symptom bother and number of patient-reported acute toxicities (as measured by the PRO-CTCAE).
EFS | From randomization until disease progression, relapse, diagnosis of a second malignant neoplasm, death or last contact, whichever occurs first, assessed up to 1 year after completion of study treatment
  Estimates of 1-year EFS for standard risk (SR) and high risk (HR) patients on each Arm MAP and Arm cabozantinib (CABO)-MAP and the corresponding 95% confidence intervals (CIs) by sex.
EFS | From randomization until disease progression, relapse, diagnosis of a second malignant neoplasm, death or last contact, whichever occurs first, assessed up to 1 year after completion of study treatment
  Estimates of 1-year EFS for SR and HR patients on each Arm MAP and Arm CABO-MAP and the corresponding 95% CIs by race.
EFS | From randomization until disease progression, relapse, diagnosis of a second malignant neoplasm, death or last contact, whichever occurs first, assessed up to 1 year after completion of study treatment
  Estimates of 1-year EFS for SR and HR patients on each Arm MAP and Arm CABO-MAP and the corresponding 95% CIs by ethnicity.

CONTACTS AND LOCATIONS:
Overall Officials: Michael W Bishop, Principal Investigator — Children's Oncology Group
Locations (183):
- United States (164):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Banner Children's at Desert, Mesa, Arizona
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Mattel Children's Hospital UCLA, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - Corewell Health Children's, Royal Oak, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Henry Ford Wyandotte Hospital, Wyandotte, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Missouri Children's Hospital, Columbia, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - UMC Cancer Center / UMC Health System, Lubbock, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (5):
  - Sydney Children's Hospital, Randwick, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Royal Children's Hospital, Parkville, Victoria
  - Perth Children's Hospital, Perth, Western Australia
- Canada (12):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - Children's Hospital, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke-Fleurimont, Sherbrooke, Quebec
  - Jim Pattison Children's Hospital, Saskatoon, Saskatchewan
  - CHU de Quebec-Centre Hospitalier de l'Universite Laval (CHUL), Québec
- New Zealand (2):
  - Starship Children's Hospital, Grafton, Auckland
  - Christchurch Hospital, Christchurch

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm